CLINICAL TRIAL: NCT02208674
Title: Early Identification and Action in CKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Alexander Chang, Clinical Investigator, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2014-0251
Record Dates: First submitted 2014-08-01; First posted 2014-08-05 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Kidney Disease; Hypertension
Keywords: chronic kidney disease; albuminuria; hypertension; dyslipidemia; cardiovascular disease; pragmatic trial; cluster randomized trial
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension; Albuminuria; Dyslipidemias; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention): Primary care provider-delivered screening and treatment for risk factors (hypertension, albuminuria, dyslipidemia) per usual care.
- Protocolized, pharmacist-delivered CKD Action Plan (Experimental): Protocolized, pharmacist-delivered screening and treatment for risk factors (hypertension, albuminuria, dyslipidemia) per KDIGO and JNC-8 recommendations.
  Interventions: Other: Protocolized, pharmacist-delivered CKD Action Plan

INTERVENTIONS:
Other: Protocolized, pharmacist-delivered CKD Action Plan — The CKD Action plan protocolizes the screening and treatment of primary risk factors for CKD progression and cardiovascular disease among individuals with stage G3A CKD
  Other Names: Health care delivery procedure
  Arms: Protocolized, pharmacist-delivered CKD Action Plan

SUMMARY:
Chronic kidney disease (CKD) is highly prevalent and associated with significantly increased risk of cardiovascular morbidity and end-stage renal disease. Evidence from randomized clinical trials suggests that treating urinary albumin excretion (UAE), dyslipidemia, and hypertension will reduce these risks. Unfortunately, less than 30% of the CKD population is screened and treated according to recommended guidelines. Using a cluster-randomized, controlled design and clinic-embedded pharmacists, this pilot pragmatic trial will randomize 6 Geisinger primary care clinics (72 patients) to usual care (group 1) or a pharmacist-directed "CKD Action Plan" (group 2). Determining the impact of the CKD Action Plan on screening and treatment guideline adherence is the primary goal of this pilot study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* eGFRCR value between 45-59 ml/min/1.73m2 in the prior 12 months
* scheduled laboratory appointment for serum creatinine testing within the next 30 days
* average systolic or diastolic blood pressure reading of at least 150 or 85 mm Hg, respectively, during the prior 12 months.

Exclusion Criteria:

* fewer than 2 blood pressure readings in the prior 12 months,
* pregnancy
* current hospitalization
* life expectancy less than 6 months as determined by the study investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Screening Urinary Albumin Excretion | At 12 months
  Completed test for urine albumin/creatinine (or urine protein/creatinine)

SECONDARY OUTCOMES:
Dyslipidemia Screening | At least once after eGFR < 60 ml/min
  One-time test for dyslipidemia (lipid panel)
ACEI or ARB Treatment if urine ACR is > 30 mg/g (diabetic) or > 300 mg/g (non-diabetic) | within 12 months of enrollment date
Statin Treatment | Within 12 months of enrollment
  If age >= 50
Blood Pressure Control-1 | Average of last two readings prior to 12 months post-enrollment
Blood Pressure--II | Average of all blood pressures within 12 month study period
Blood Pressure--III | at 12 months post enrollment
  Target blood pressure attained (using KDIGO criteria) based on average of last 2 clinic readings within 12 month study period
Biochemical Surveillance | two weeks after initiation or titration of ACEI or ARB
  Test order for serum creatinine, potassium, and sodium within two weeks of ACEI or ARB initiation or titration.
Symptomatic Adverse Drug Event | At 12 months post-enrollment
  Angioedema, anaphylaxis, syncope, hypotension, or myopathy after initiation or titration of antihypertensive and/or statin drug
Patient and Provider Satisfaction | 9-12 months post study start date
  Based on administered surveys
Cystatin C Supplementary Screening | within 12 months of enrollment date
  One-time serum cystatin C test for individuals with eGFR between 45 and 59 ml/min and urine albumin-creatinine < 30 mg/g.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Chang, MD, MS, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Health System, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Data for this study may be obtained upon request, after permission to do so is granted by the Geisinger IRB and information security office. Readers should contact the principal investigator (achang@geisinger.edu) for further information.

REFERENCES:
- [Background] Chang AR, Evans M, Yule C, Bohn L, Young A, Lewis M, Graboski E, Gerdy B, Ehmann W, Brady J, Lawrence L, Antunes N, Green J, Snyder S, Kirchner HL, Grams M, Perkins R. Using pharmacists to improve risk stratification and management of stage 3A chronic kidney disease: a feasibility study. BMC Nephrol. 2016 Nov 8;17(1):168. doi: 10.1186/s12882-016-0383-7. PMID 27825313
- See also: Related Info — https://bmcnephrol.biomedcentral.com/articles/10.1186/s12882-016-0383-7